CLINICAL TRIAL: NCT02777424
Title: Prothrombin Complex Concentrate Versus Fresh Frozen Plasma to Correct Coagulation Disorders in Adult Neurosurgical Patients
Brief Title: CPP Versus PFC to Correct Coagulation Disorders in Adult Neurosurgical Patients
Acronym: CLOT-CRANE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGR_2014-22
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Factor IX

ARMS (2):
- Prothrombin Complex Concentrate (Experimental): Administration of a single dose of prothrombin complex concentrate (25 U/kg equivalent factor IX)
  Interventions: Drug: Prothrombin Complex Concentrate
- Fresh Frozen Plasma (Active Comparator): Administration of a single dose of fresh frozen plasma of 15 mL/kg
  Interventions: Biological: Fresh Frozen Plasma

INTERVENTIONS:
Drug: Prothrombin Complex Concentrate — Non-activated prothrombin complex concentrate containing factors II, VII, IX and X and proteins C & S
  Arms: Prothrombin Complex Concentrate
Biological: Fresh Frozen Plasma — Pooled collection of plasma from donors
  Arms: Fresh Frozen Plasma

SUMMARY:
This prospective, randomized, multicenter study is performed to determine whether prothrombin complex concentrates confers any benefits over fresh frozen plasma in adult neurological patients with coagulation disorders (PT value less than 60%).

DETAILED DESCRIPTION:
The coagulation disorders increase the risk of bleeding and are a risk factor of intracranial hemorrhagic complications in neurosurgical patients. They are diagnosed more often in emergency on a PT value less than 60% and so they should be corrected as soon as possible. Two therapeutic strategies are proposed by French or international recommendations: transfusion of fresh frozen plasma (FFP) or administration of prothrombin complex concentrates (PCC).

This prospective, randomized, multicenter study with blinded assessment of the primary endpoint, is performed to determine whether PCC confers any benefits over FFP in the neurological patients with coagulation disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient with spontaneous intracranial hemorrhage or traumatic intracranial hemorrhage or patient requiring neurological surgery
* Coagulation disorder defined by PT less than 60%

Exclusion Criteria:

* Concomitant use with oral anticoagulant drugs
* Acquired deficiency of coagulation factors whose treatment is established
* Hypersensitivity to a PCC
* History of thrombocytopenia induced by heparin
* Disseminated intravascular coagulation
* Extracranial active bleeding
* Hypersensitivity to vitamin K

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with correction of prothrombin time (PT more than 60%) | End of treatment administration (an average of 1 hour)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Lille, Lille
  - CHU de NANCY, Nancy
  - Fondation Ophtalmologique Adolphe de Rothschild (FOR), Paris
  - Hôpital Foch, Suresnes

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112